CLINICAL TRIAL: NCT01578122
Title: Evaluation of the Efficacy of Elastic Compression in Preventing Post-thrombotic Syndrome. Randomised Non-inferiority Study for Ankle Pressure Targeted at 25 mm Hg Versus 35 mm Hg
Brief Title: Elastic Compression Stockings for Prevention of Post-thrombotic Syndrome
Acronym: CELEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Innothera (Industry)
Collaborators: University Hospital, Grenoble (Other); Floralis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVE301-10 (Themas) : DCIC/1028; 2010-A01078-31 (Other: French Agency for the Safety of Health Care Products)
Record Dates: First submitted 2012-04-13; First posted 2012-04-16 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2019-08

CONDITIONS: Deep Vein Thrombosis; Post-thrombotic Syndrome
Keywords: post-thrombotic syndrome; prevention; deep vein thrombosis; elastic compression stockings; compliance; quality of life
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome; Patient Compliance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 25mmHg ECS (Experimental): Thigh-length graduated elastic compression stockings applying 25mmhg of targeted pressure at the ankle worn daily for two years
  Interventions: Device: 25mmHg ECS
- 35mmHg ECS (Active Comparator): Thigh-length graduated elastic compression stockings applying 35 mmhg of targeted pressure at the ankle worn daily for two years
  Interventions: Device: 35 mmHg ECS

INTERVENTIONS:
Device: 25mmHg ECS — Thigh-length graduated elastic compression stockings applying 25 mmhg of targeted pressure at the ankle worn daily (from morning to night) for two years.
  Before receiving the randomly allocated treatment, each patient will wear cotton, class III Varisma Comfort® stay-up stockings (20-36 mm Hg).
  Other Names: ACTYS 25® for women; LEGGER 25® for men
  Arms: 25mmHg ECS
Device: 35 mmHg ECS — Thigh-length graduated elastic compression stockings applying 35mmhg of pressure at the ankle worn daily (from morning to night) for two years Before receiving the randomly allocated treatment, each patient will wear cotton, class III Varisma Comfort® stay-up stockings (20-36 mm Hg).
  Other Names: ACTYS 35® for women; LEGGER 35® for men
  Arms: 35mmHg ECS

SUMMARY:
Post thrombotic syndrome (PTS) is a frequent and burdensome complication of proximal deep-vein thrombosis.Therapeutic options for PTS are limited and mainly rely on its prevention. Therapeutic trials evidenced that elastic compression stockings (ECS) applying 30-40mmHg of pressure at the ankle reduced the rate of PTS by 50%. Although ECS are unlikely to cause harm, in clinical practice, compliance to this treatment appears to be low as ECS may be difficult to apply and to wear.

ECS with a lighter compression strength (20-30mmHg) might be easier to apply and be more comfortable. This could favor a better compliance.

CELEST is a randomized, multicentre, double-blind trial which aims to determine whether ECS applying 25mmHg of targeted pressure at the ankle are non inferior to ECS applying 35mmHg of targeted pressure at the ankle

DETAILED DESCRIPTION:
CELEST trial is a controlled, randomized, multicentre, non-inferiority double-blind trial which aims to determine whether ECS applying 25mmHg of targeted pressure at the ankle are non inferior to ECS applying 35mmHg of targeted pressure at the ankle. Patients with a first acute symptomatic proximal DVT will be randomized to wear for two years either ECS applying 25mmHg of targeted pressure at the ankle or ECS applying 35mmHg of targeted pressure at the ankle. All patients will be prescribed anticoagulants for at least three months. The primary outcome will be the rate of PTS assessed with the Villalta scale in both arms of the study during the 2 years study period. Rate of compliance,severity of PTS and quality of life in both groups will constitute the main secondary outcomes.

ELIGIBILITY:
Inclusion criteria

* Patient (male/female) at least 18 years old
* Patient presenting with an initial episode of proximal deep vein thrombosis (DVT) confirmed by an additional examination (echo-Doppler scan) taken no more than 8 days previously :

the proximal character defined by a DVT from the collecting trunk extending from the tibial-peroneal trunk to the inferior vena cava inclusive the unilateral character concerns only the proximal part. Patients with a distal DVT on the contralateral member the day of diagnosis can be included The notion of initial episode concerns only the proximal part. Patients with a preceding DVT limited to distal part can be included

* with no trophic disorders at baseline (CEAP class 4, 5 or 6 excluded)
* with or without pulmonary embolism
* Patient capable of benefiting from anticoagulant therapy of at least 3 months duration
* Available to participate in a clinical trial with a 24-month follow-up period and for which a delivery of study products may be possible throughout its participation (delivery possible only in Metropolitan France)
* Life expectancy greater than 24 months
* Volunteer to take part in the study, having signed the consent form after receiving sufficient information and the information leaflet
* Person affiliated to social security or the recipient of a similar scheme.

non inclusion criteria

* Patients with at least one of these contraindications to compression treatment:

  * phlegmasia cerulea dolens,
  * septic thrombosis,
  * product intolerance, allergic reaction to one of the components
  * Arteritis obliterans stage III and IV of the lower limbs (IPS<0.6),
  * Micro-angiopathy, advanced diabetes,
  * Decompensated heart failure,
  * Skin infections: anti-infective treatment must precede compression therapy,
  * Weeping skin diseases of the leg.
  * Compression treatment technically impossible during the study
* Patients presenting with bilateral venous thrombosis of the lower limbs.
* Patient having received fibrinolytic treatment, mechanical thrombo-aspiration or venous repermeation surgery for venous thrombosis justifying inclusion
* Patients having undergone mechanical interruption of the inferior vena cava.
* Patients for whom long-term elastic compression for the treatment of lymphatic venous insufficiency (patients with lymphoedema), for instance, is indicated prior to DVT. Patients with elastic compression for primary thromboprophylaxis of thromboembolic disease (TED) are eligible.
* Patients presenting with oedema unrelated to venous insufficiency or in whom oedema is likely to develop within 2 years.
* Patients receiving diuretic treatment for more than 3 months due to heart failure.
* Pregnant women
* Person deprived of liberty by a legal or administrative decision, person under legal protection.
* Patient currently participating in a clinical trial or having taken part in a clinical trial in the month preceding inclusion
* Patient presenting with a history of mental or psychiatric illness or any other factor restricting his/her ability to participate in an informed manner and in compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2012-06-29 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
To show that elastic compression with ankle pressure targeted at 25 mm Hg is not inferior in preventing the onset of clinical post-thrombotic syndrome to a target ankle pressure of 35 mm Hg (recommended pressure being greater than 30 mm Hg) | 24 months
  cumulative incidence 24 months after inclusion of PTS apparition defined by the Villalta score > or equal to 5. A visual guide will be given to investigators to assist them and standardize PTS evaluation. Investigators will receive a Villalta training during set up visits.

SECONDARY OUTCOMES:
superiority of targeted pressure at 35 mm Hg for compliant patients. Analysis of the primary endpoint per protocol amongst patients responding to the definition of compliance for compression scheduled by randomization | 24 months
  analysis of primary endpoint (cumulative incidence of PTS) amongst patients responding to the definition of observance for compression scheduled by randomization. It means a per protocol analysis. The per protocol analysis defined as follow : patients ideally compliant (see next secondary outcome measure with self declaration of compression carrying superior or equal to 80 % especially)and patients with respect to randomization.
Superiority of 25 mm Hg on the therapeutic compliance criterion | 24 months
  Superiority of 25 mm Hg on the therapeutic compliance criterion at 24 months
  Compliance is defined by 2 conditions :
  1. Girerd adapted to elastic compression stocking score adjusted between 0 and 2 (the question 2 will not be taken into account beacause not adapted to the logistics of the study)
  2. because of French clinical practices it should be pertinent to take into consideration 2 compliance type :
     1. ideal compliance : Self declaration ≥ 80 % (reference PRANDONI)
     2. adequate compliance : self declaration between 50 and 79% for (French references Delluc and Optimev study)
superiority of 25 mm Hg for constraints related to compression and chronic venous insufficiency quality of life (CIVIQ) | 3 months, 12 months, 24 months
  CIVIQ quality of life (CIVIQ 20) specific to chronic venous insufficiency at 3 months, 12 months and 24 months and questionnaire about constraints of compression stockings.
non inferiority of 25 mm Hg for the comparative evaluation of the symptomatic effect of short-term compression (pain, sensation of oedema) form baseline to 3 months | 3 months
  Comparison of evolution at short-term (3 months) of venous thrombosis symptoms (pain, oedema feeling). Self assessment by VAS of pain and oedema feeling once a week during 3 months. Assessment by the investigator at inclusion and during visit at 3 months (ankle measurement, clinical signs) will be done also. A statistical analysis will be done as soon as 3 months follow up data will be verified to evaluate symptoms evolution due to deep venous thrombosis.
Non-inferiority of 25 mm Hg for changes in overall quality of life evaluated on the basis of the EUROQUOL questionnaire | 3months, 12 months, 24 months
  Non-inferiority of 25 mm Hg for changes in overall quality of life evaluated on the basis of the EUROQUOL questionnaire (EQ5D)
non inferiority of 25 mm Hg for the intensity of long term chronic venous insufficiency symptoms (12 months and 24 months) | 12 and 24 months
  Long term assessment of evolution and intensity of symptoms (pain, oedema feeling) related to potential post-thrombotic syndrome apparition
  * Monthly self-assessment by VAS for pain and oedema feeling during 24 months. It will be done at the end of each month and will focus on symptoms intensity (last week of the month)
  * An assessment will be done by investigator, in addition of previous criterion, at 12 and 24 months
  * Assessment with the Ginsberg score (interview by the investigator at 12 and 24 months)
  * Comparison of averages on Villalta score (quantitative)
non inferiority of 25 mm Hg for the onset of permanent trophic disorders | 3 months, 12 and 24 months
  CEAP classification evaluated by investigator at 3, 12 and 24 months
non inferiority of 25 mm Hg for the onset of sequalae or post thrombotic residues on an duplex scan at 3 months, 12 and 24 months | 3, 12 and 24 months
  Assessment by duplex scan of deep and superficial veins at 3, 12 and 24 months
  * Assessment by duplex scan of deep reflux (>1s in femoral vein, and/or popliteal vein, tibio peroneal trunck)
  * Assessment by duplex scan of superficial reflux (> 0.5s in great saphenous vein, small saphenous vein, perforating veins)
  * Assessment by echographic score of thickness and location of residual thrombus
  * Assessment by duplex scan of re-canalization of collectors trunks and/or parietal sequalae
testing for the prognostic factors of the onset post thrombotic syndrome and comparison of the onset kinetics of post thrombotic syndrome | 24 months
  variables tested as prognostic factors of post thrombotic syndrome apparition :
  * location of the upper pole of thrombus
  * kinetic of thrombus lysis by duplex scan at 3 months
  * Idiopathic nature of TED
  * Delay of diagnostic of deep venous thrombosis
  * Initial intensity of deep venous thrombosis symptoms
  * Initial evolution of symptoms of deep venous thrombosis between J0 and 3 months
  * Persistence of the symptoms at 3 months
  * Patient's characteristics
  * Kinetic of of Villalta score apparition ≥ 5 by survival curve
  * Kinetic of post thrombotic syndrome apparition by Villalta score
test for key factors in good compliance | 24 months
  Compliance evaluation according to the 2 axes defined on third outcome measure and research of determinants of good compliance by specific questionnaire
Adverse events | 24 months
  description and comparison of the incidence of adverse events including unexpected adverse events, events expected with this type of disease (recurrence of the venous thromboembolic disease, recurrence of deep vein thrombosis, pulmonary embolism, superficial venous thrombosis, venous ulcer) and events possibly related to the study treatment (arterial decompensation passing to Lerich stage III or IV, skin intolerance)
Subgroups analysis of the primary objective and secondary objectives according to the gender stratification criterion and age | 24 months
  Stratification on age (more or less than 65 years-old) for testing the hypothesis by subgroups analysis of the benefit of a better adaptation of compression 25 mm Hg on older subjects, as suggested by S. Khan.
superiority of 25 mmHg on 35 mmHg in preventing the onset of clinical post thrombotic syndrome | 24 months
  superiority of 25 mmHg on 35 mmHg in preventing the onset of clinical post thrombotic syndrome. Outcome measure identical to primary endpoint
sensitivity analysis of primary endpoint excluding patients with a differential diagnosis can explain a Villalta score ≥ 5 | 24 months
  sensitivity analysis of primary endpoint excluding patients with a differential diagnosis which could explain a Villalta score ≥ 5. Outcome measure identical to primary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc BOSSON, MD, PhD, Principal Investigator — CIC Grenoble
Locations (57):
- France (57):
  - Cabinet, Lyon, Rhônes Alpes
  - Cabinet, Aix-les-Bains
  - Cabinet, Alençon
  - Clinique Victor PAUCHET, Amiens
  - CHRU Amiens, Amiens
  - Cabinet, Amiens
  - Chu Angers, Angers
  - Cabinet, Annecy
  - Chra Annecy, Annecy
  - Centre Hospitalier d'Armentieres, Armentières
  - CH Armentières, Armentières
  - Cabinet, Bordeaux
  - Cabinet, Bourgoin
  - Ch Bourgoin-Jallieu, Bourgoin
  - Hia Brest, Brest
  - Chu Brest, Brest
  - CHU, Caen
  - Cabinet, Carcassonne
  - Cabinet, Chalon-sur-Saône
  - Ch Chalon Sur Saone, Chalon-sur-Saône
  - CH de Chambéry, Chambéry
  - Cabinet, Clapiers
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Cabinet, Dijon
  - Hôpital du bocage, Dijon
  - Cabinet, Échirolles
  - Cabinet, Genas
  - Cabinet, Grenoble
  - Chu Grenoble, Grenoble
  - Cabinet, Hennebont
  - Cabinet, Issy-les-Moulineaux
  - Ch La Rochelle, La Rochelle
  - Cabinet, Lille
  - Chru Lille, Lille
  - Hopital Saint Philibert, Lomme
  - CH Pierre-Bénite, Lyon
  - CH Mâcon, Mâcon
  - Cabinet, Montbonnot-Saint-Martin
  - Cabinet, Montélimar
  - Cabinet, Montigny-lès-Metz
  - Cabinet, Montluçon
  - Chu Montpellier, Montpellier
  - Chu Hotel Dieu, Nantes
  - CHR Orléans, Orléans
  - HEGP, Paris
  - Hôpital St Joseph, Paris
  - Cabinet, Péronne
  - Cabinet, Saint-Alban
  - Cabinet, Saint-Aubin-sur-Scie
  - Chu St Etienne, Saint-Etienne
  - Cabinet, Sélestat
  - Cabinet, Thonon-les-Bains
  - Chu Toulouse, Toulouse
  - Cabinet, Tournefeuille
  - Cabinet, Villeurbanne
  - Cabinet, Vizille

REFERENCES:
- [Background] Fowkes FJ, Price JF, Fowkes FG. Incidence of diagnosed deep vein thrombosis in the general population: systematic review. Eur J Vasc Endovasc Surg. 2003 Jan;25(1):1-5. doi: 10.1053/ejvs.2002.1778. PMID 12525804
- [Background] Oger E. Incidence of venous thromboembolism: a community-based study in Western France. EPI-GETBP Study Group. Groupe d'Etude de la Thrombose de Bretagne Occidentale. Thromb Haemost. 2000 May;83(5):657-60. PMID 10823257
- [Background] Prandoni P, Kahn SR. Post-thrombotic syndrome: prevalence, prognostication and need for progress. Br J Haematol. 2009 May;145(3):286-95. doi: 10.1111/j.1365-2141.2009.07601.x. Epub 2009 Feb 13. PMID 19222476
- [Background] Prandoni P, Lensing AW, Cogo A, Cuppini S, Villalta S, Carta M, Cattelan AM, Polistena P, Bernardi E, Prins MH. The long-term clinical course of acute deep venous thrombosis. Ann Intern Med. 1996 Jul 1;125(1):1-7. doi: 10.7326/0003-4819-125-1-199607010-00001. PMID 8644983
- [Background] Prandoni P, Villalta S, Bagatella P, Rossi L, Marchiori A, Piccioli A, Bernardi E, Girolami B, Simioni P, Girolami A. The clinical course of deep-vein thrombosis. Prospective long-term follow-up of 528 symptomatic patients. Haematologica. 1997 Jul-Aug;82(4):423-8. PMID 9299855
- [Background] Gabriel F, Labios M, Portoles O, Guillen M, Corella D, Frances F, Martinez M, Gil J, Saiz C. Incidence of post-thrombotic syndrome and its association with various risk factors in a cohort of Spanish patients after one year of follow-up following acute deep venous thrombosis. Thromb Haemost. 2004 Aug;92(2):328-36. doi: 10.1160/TH03-11-0700. PMID 15269829
- [Background] Kahn SR, Ginsberg JS. Relationship between deep venous thrombosis and the postthrombotic syndrome. Arch Intern Med. 2004 Jan 12;164(1):17-26. doi: 10.1001/archinte.164.1.17. PMID 14718318
- [Background] Kahn SR, Hirsch A, Shrier I. Effect of postthrombotic syndrome on health-related quality of life after deep venous thrombosis. Arch Intern Med. 2002 May 27;162(10):1144-8. doi: 10.1001/archinte.162.10.1144. PMID 12020185
- [Background] Bergqvist D, Jendteg S, Johansen L, Persson U, Odegaard K. Cost of long-term complications of deep venous thrombosis of the lower extremities: an analysis of a defined patient population in Sweden. Ann Intern Med. 1997 Mar 15;126(6):454-7. doi: 10.7326/0003-4819-126-6-199703150-00006. PMID 9072931
- [Background] Brandjes DP, Buller HR, Heijboer H, Huisman MV, de Rijk M, Jagt H, ten Cate JW. Randomised trial of effect of compression stockings in patients with symptomatic proximal-vein thrombosis. Lancet. 1997 Mar 15;349(9054):759-62. doi: 10.1016/S0140-6736(96)12215-7. PMID 9074574
- [Background] Prandoni P, Lensing AW, Prins MH, Frulla M, Marchiori A, Bernardi E, Tormene D, Mosena L, Pagnan A, Girolami A. Below-knee elastic compression stockings to prevent the post-thrombotic syndrome: a randomized, controlled trial. Ann Intern Med. 2004 Aug 17;141(4):249-56. doi: 10.7326/0003-4819-141-4-200408170-00004. PMID 15313740
- [Background] Milne AA, Ruckley CV. The clinical course of patients following extensive deep venous thrombosis. Eur J Vasc Surg. 1994 Jan;8(1):56-9. doi: 10.1016/s0950-821x(05)80121-5. PMID 8307217
- [Background] Partsch H, Blattler W. Compression and walking versus bed rest in the treatment of proximal deep venous thrombosis with low molecular weight heparin. J Vasc Surg. 2000 Nov;32(5):861-9. doi: 10.1067/mva.2000.110352. PMID 11054217
- [Background] Kahn SR, Elman E, Rodger MA, Wells PS. Use of elastic compression stockings after deep venous thrombosis: a comparison of practices and perceptions of thrombosis physicians and patients. J Thromb Haemost. 2003 Mar;1(3):500-6. doi: 10.1046/j.1538-7836.2003.00098.x. PMID 12871457
- [Background] Benko T, Cooke EA, McNally MA, Mollan RA. Graduated compression stockings: knee length or thigh length. Clin Orthop Relat Res. 2001 Feb;(383):197-203. PMID 11210954
- [Background] Sajid MS, Tai NR, Goli G, Morris RW, Baker DM, Hamilton G. Knee versus thigh length graduated compression stockings for prevention of deep venous thrombosis: a systematic review. Eur J Vasc Endovasc Surg. 2006 Dec;32(6):730-6. doi: 10.1016/j.ejvs.2006.06.021. Epub 2006 Aug 23. PMID 16931066
- [Background] Nelson EA, Harper DR, Prescott RJ, Gibson B, Brown D, Ruckley CV. Prevention of recurrence of venous ulceration: randomized controlled trial of class 2 and class 3 elastic compression. J Vasc Surg. 2006 Oct;44(4):803-8. doi: 10.1016/j.jvs.2006.05.051. PMID 17012004
- [Background] Arpaia G, Cimminiello C, Mastrogiacomo O, de Gaudenzi E. Efficacy of elastic compression stockings used early or after resolution of the edema on recanalization after deep venous thrombosis: the COM.PRE Trial. Blood Coagul Fibrinolysis. 2007 Mar;18(2):131-7. doi: 10.1097/MBC.0b013e328011f2dd. PMID 17287629
- [Background] Roumen-Klappe EM, den Heijer M, van Rossum J, Wollersheim H, van der Vleuten C, Thien T, Janssen MC. Multilayer compression bandaging in the acute phase of deep-vein thrombosis has no effect on the development of the post-thrombotic syndrome. J Thromb Thrombolysis. 2009 May;27(4):400-5. doi: 10.1007/s11239-008-0229-7. Epub 2008 May 15. PMID 18480967
- [Background] Delluc A, Gouedard C, De Saint Martin L, Garcia C, Roguedas AM, Bressollette L, Misery L, Mottier D, Le Gal G. [Incidence, risk factors and skin manifestations of post-thrombotic syndrome: a four-year follow-up of patients included in the EDITH study]. Rev Med Interne. 2010 Nov;31(11):729-34. doi: 10.1016/j.revmed.2010.07.018. Epub 2010 Sep 29. French. PMID 20880613
- [Derived] Galanaud JP, Genty-Vermorel C, Barrellier MT, Becker F, Jabbour V, Blaise S, Bura-Riviere A, Comte A, Grange C, Guenneguez H, Maufus M, Ouvry P, Richaud C, Rolland C, Schmidt J, Sevestre MA, Verriere F, Bosson JL; CELEST trial investigators. 25 mm Hg versus 35 mm Hg elastic compression stockings to prevent post-thrombotic syndrome after deep vein thrombosis (CELEST): a randomised, double-blind, non-inferiority trial. Lancet Haematol. 2022 Dec;9(12):e886-e896. doi: 10.1016/S2352-3026(22)00247-2. PMID 36455606